CLINICAL TRIAL: NCT00850057
Title: A Phase 1, Open Label, Dose-escalation, Pharmacodynamic Study of Intranodal Injection of Adenovirus-CD154 (Ad-ISF35) in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Pharmacodynamic (PD) Study of Intranodal Adenovirus-CD154 (Ad-ISF35) in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Memgen, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD-060201; NCT00783874 (obsolete NCT alias)
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Intranodal injection of Ad-ISF35 — Ad-ISF35, a replication-defective recombinant type V adenovirus encoding a recombinant humanized CD154 homolog (ISF35).

SUMMARY:
Primary Objectives

* To determine the safety and maximum tolerated dose (MTD) of Adenovirus-CD154 (Ad-ISF35) when it is injected directly into the lymph nodes of patients with CLL or SLL.

Secondary Objectives

* To determine and monitor clinical and biological responses in patients treated with injections of Ad-ISF35.
* To determine how ISF35 works in CLL/SLL patients' cells.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of B-cell CLL/SLL including

   * Lymphocytosis of monoclonal B-cells co-expressing ≥ one B-cell marker (CD19, CD20, or CD23) and CD5 in peripheral blood or lymph node AND
   * Bone marrow with ≥ 30% mononuclear cells having the CLL/SLL phenotype.
2. Presence of at least ONE single accessible AND palpable lymph node in the cervical, supraclavicular, axillary, or inguinal regions. The size of the lymph nodes must be larger than 2x2 cm in the horizontal and perpendicular axes.
3. Intermediate or High risk, poor prognosis CLL/SLL
4. Indication for treatment as defined by the NCI Working Group Guidelines:

   * Massive (i.e. > 6 cm below the left costal margin) or progressive splenomegaly OR
   * Massive lymph nodes or nodal clusters (i.e. > 10 cm in longest diameter), or progressive lymphadenopathy OR
   * Grade 2 or 3 fatigue OR
   * Fever ≥ 100.5˚F or night sweats for greater than 2 weeks without documented infection OR
   * Presence of weight loss ≥ 10% over the preceding 6 months OR
   * Progressive lymphocytosis with an increase of ≥ 50% over a 2-month period or an anticipated doubling time of less than 6 months.
   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and / or thrombocytopenia.
   * Autoimmune anemia and / or thrombocytopenia poorly responsive to corticosteroid therapy.
5. Males and females 18 years of age and older
6. Laboratory parameters as specified below:

   * Hematologic: Hemoglobin ≥ 10 g/dL (may be post-transfusion); platelet count ≥ 50 x103/mm3
   * Hepatic: Total Bilirubin < 2 X ULN, and ALT and AST < 2 x ULN
   * Renal: Creatinine ≤ 2 X ULN
7. ECOG Performance Status ≤ 2
8. Anticipated survival of at least 3 months
9. For men and women of child-producing potential, use of effective barrier contraceptive methods during the study and for one month following treatment.
10. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
11. Negative test results for current/active infection with HIV-1, HIV-2, HTLV-1, HTLV-2, hepatitis A, B, C within 30 days of registration. (Antibody, antigen and nucleic acid tests acceptable, depending on institutional standards.).

Exclusion Criteria:

1. Pregnant or nursing women
2. Treatment with chemotherapy or monoclonal antibody within 28 days prior to entering the study.
3. Treatment with chemotherapy or monoclonal antibody during the time of participation in this trial.
4. Grade 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
5. Severe or debilitating pulmonary disease (dyspnea at rest, significant shortness of breath, COPD)
6. Participation in any investigational drug study within 28 days prior to ISF35 administration. (Patient must have recovered from all acute effects of previously administered investigational agents)
7. History of malignancy other than CLL within five years of registration, except patients with adequately treated basal, squamous cell carcinoma or localized cervical cancer.
8. Active symptomatic fungal, bacterial and/or viral infection including active HIV or viral (A, B or C) hepatitis.
9. Any illness or condition that in the opinion of the Investigator may affect safety of treatment or evaluation of any the study's endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Determine the safety and maximum tolerated dose (MTD) of Adenovirus-CD154 (Ad-ISF35) when injected directly into lymph nodes of patients with CLL/SLL. | 2 years

SECONDARY OUTCOMES:
Determine and monitor clinical and biological responses in patients treated with intranodal injections of Ad-ISF35. | 2 years
Determine pharmacodynamic (PD) parameters in patients treated with intranodal injections of ISF35. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Januario Castro, M.D., Principal Investigator — Assistant Clinical Professor in the Blood and Marrow Transplantation Division
Locations (1):
- University of California, San Diego Moores Cancer Center, La Jolla, California, United States